CLINICAL TRIAL: NCT01134471
Title: Improvement of Hemostasis Techniques After Median Sternotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Aarhus University Hospital (Other)
Collaborators: Ceremed, Inc. (Industry)
Responsible Party: Rikke Vestergaard/ MD, Aarhus University Hospital, Skejby, Cardiothorasic surgery dept.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ostene-project
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Sternal Dehiscence; Sternal Infection; Sternal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention)
- Bonewax (Active Comparator): Patients treated with the hemostatic bonewax
  Interventions: Device: Bonewax
- Ostene (Active Comparator): Patients treated with the hemostatic Ostene
  Interventions: Device: Ostene

INTERVENTIONS:
Device: Ostene — applied to sternal surface
  Arms: Ostene
Device: Bonewax — applied to sternal surface
  Arms: Bonewax

SUMMARY:
The purpose of this study is to compare 2 different hemostatic agents (Bonewax and Ostene)to a control group with regards to bleeding, bone healing, pain and infection in a patient group all undergoing median sternotomy.

ELIGIBILITY:
Inclusion Criteria:

* men undergoing elective cardiac surgery at the Cardiac surgery department of Aarhus University Hospital, Skejby
* no clopidogrel-treatment
* no osteoporoses
* less than 2 co-morbidities in the form of obesity (BMI>30), COPD, chronic steroid use, renal failure, immunosuppression and diabetes

Exclusion Criteria:

* profuse sternal bleeding
* serious complications to the surgery fx cerebral infarction
* re-operation due to bleeding

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Bone healing in sternum | 6 months after surgery
Questionnaire regarding physical and emotional well being | 6 months after surgery
Pain-score (VAS) | 6 months

SECONDARY OUTCOMES:
Blood product consumption | 6 months
Mediastinitis | 6 months
superficial infection | 6 months
Bleeding through the chest tube | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Vestergaard, MD, Principal Investigator — Dept. of Cardiothoracic surgery, Aarhus University Hospital, Skejby
Locations (1):
- Aarhus University Hospital, Skejby, Dept. of Cardiothoracic surgery, Aarhus, Denmark